CLINICAL TRIAL: NCT03775070
Title: An Open Label, Single-armed, Exploratory Study of Simvastatin Therapy on the Cardiac Function in Patients With Dilated Cardiomyopathy.
Brief Title: Simvastatin Therapy in Patients With Dilated Cardiomyopathy.
Acronym: SavDCM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201806014MINB
Record Dates: First submitted 2018-12-03; First posted 2018-12-13 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Simvastatin (Experimental): Simvastatin, 0.5mg/kg/d(maximum 20mg), once daily
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — * Starting dosage: in adult, the dose of simvastatin is 10 mg once daily. In children, the dose is 0.25mg/Kg/day (maximum dose: 10 mg/d).
  * Target dosage: in adult, the dose of simvastatin is 20 mg once daily. In children, the dose is 0.5mg/Kg/day (maximum dose: 20 mg/d).
  * The basic anti-congestive medication will be kept as the same.
  * The dosage may be titrated to a lesser dose by investigators according to the patient's condition.

SUMMARY:
Dilated cardiomyopathy (DCM) is the most common childhood cardiomyopathy and is associated with significant early morbidity and mortality. About half of patients die or require heart transplantation within 5 years of diagnosis. The medical therapy for DCM with heart failure includes anti-congestive medications and antiplatelet therapy. Those who fail to improve within the first year of diagnosis usually deteriorated even upon aggressive anti-congestive medications. The investigators had conducted precision-medicine-based approach to provide strategic approach as drug repurposing to identify new treatments. The investigators have identified the beneficial effects from a statin, simvastatin, to restore the cardiac contractility. The investigators would further assess the efficacy of simvastatin to improve the cardiac function in patients with DCM.

DETAILED DESCRIPTION:
Dilated cardiomyopathy (DCM) is the most common childhood cardiomyopathy and is associated with significant early morbidity and mortality. About half of patients die or require heart transplantation within 5 years of diagnosis. The survival advantage from transplantation is limited, particularly in DCM infants.

The medical therapy for DCM with heart failure includes anti-congestive medications and antiplatelet therapy. Those who fail to improve within the first year of diagnosis usually deteriorated even upon aggressive anti-congestive medications. The investigators had conducted precision-medicine-based approach to provide strategic approach as drug repurposing to identify new treatments. The investigators have identified the beneficial effects from a statin, simvastatin, to restore the cardiac contractility in a DCM proband.The initial experience in the proband is promising.

Simvastatin is effective in lowing LDL and cholesterol, thereby to improve the outcome of patients with coronary arterial disease, familiar hypercholesterolemia, etc. For children, though the dosage range and the indication remain unclear, it had been used in children with various diseases. Simvastatin had been given in a small cohort of adult DCM. Patients treated with simvastatin had a lower New York Heart Association functional class compared with those receiving placebo. The LVEF also improved in the simvastatin group. The investigators would further assess the efficacy of simvastatin to improve the cardiac function in patients with DCM.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have already received anti-congestive medications for at least three months and still have compromised LV function (LVEF < 45% and the Z score of the LV end-diastolic diameter > 2.0).
* Patients who have persistent or even worsening heart failure after one month of anti-congestive medications.
* Patients who have positive family history of dilated cardiomyopathy and have received anti-congestive medications for one week.

Exclusion Criteria:

* Patients who underwent prior cardiac surgery. Those who received DCM related cardiac surgery, such as mitral valve plasty, for longer than a year are not subject to this restriction.
* Patients who had liver / renal dysfunction.
* Patients who are pregnant or plan to pregnancy in the period of study.
* Patients who are intolerance to simvastatin therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change from base line in left ventricular ejection fraction and end-diastolic dimention by cardiac ultrasound. | baseline, 1st month(The 1st month follow-up time tolerates a 0.5-month window )
Change from base line in left ventricular ejection fraction and end-diastolic dimention by cardiac ultrasound. | baseline, 3rd month(The 3rd month follow-up time tolerates a 1-month window )
Change from base line in left ventricular ejection fraction and end-diastolic dimention by cardiac ultrasound. | baseline, 6th month(The 6th month follow-up time tolerates a 1-month window )
Change from base line in left ventricular ejection fraction and end-diastolic dimention by cardiac ultrasound. | baseline, 9th month(The 9th month follow-up time tolerates a 1-month window )
Change from base line in left ventricular ejection fraction and end-diastolic dimention by cardiac ultrasound. | baseline, 12th month(The 12th month follow-up time tolerates a 1-month window )
Change from base line in left ventricular ejection fraction and end-diastolic dimention by cardiac ultrasound. | baseline, 15th month(The 15th month follow-up time tolerates a 1-month window )
Change from base line in left ventricular ejection fraction and end-diastolic dimention by cardiac ultrasound. | baseline, 18th month(The 18th month follow-up time tolerates a 1-month window )
Change from base line in left ventricular ejection fraction and end-diastolic dimention by cardiac ultrasound. | baseline, 21st month(The 21th month follow-up time tolerates a 1-month window )
Change from base line in left ventricular ejection fraction and end-diastolic dimention by cardiac ultrasound. | baseline, 24th month(The 24th month follow-up time tolerates a 1-month window )
Change from baseline in N-terminal pro-brain natriuretic peptide level.natriuretic peptide level. | baseline, 3rd month(The 3rd month follow-up time tolerates a 1-month window )
Change from baseline in N-terminal pro-brain natriuretic peptide level.natriuretic peptide level. | baseline, 6th month(The 6th month follow-up time tolerates a 1-month window )
Change from baseline in N-terminal pro-brain natriuretic peptide level.natriuretic peptide level. | baseline, 9th month(The 9th month follow-up time tolerates a 1-month window )
Change from baseline in N-terminal pro-brain natriuretic peptide level.natriuretic peptide level. | baseline, 12th month(The 12th month follow-up time tolerates a 1-month window )
Change from baseline in N-terminal pro-brain natriuretic peptide level.natriuretic peptide level. | baseline, 15th month(The 15th month follow-up time tolerates a 1-month window )
Change from baseline in N-terminal pro-brain natriuretic peptide level.natriuretic peptide level. | baseline, 18th month(The 18th month follow-up time tolerates a 1-month window )
Change from baseline in N-terminal pro-brain natriuretic peptide level.natriuretic peptide level. | baseline, 21st month(The 21th month follow-up time tolerates a 1-month window )
Change from baseline in N-terminal pro-brain natriuretic peptide level.natriuretic peptide level. | baseline, 24th month(The 24th month follow-up time tolerates a 1-month window )

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v3.0 | Up to 24 months
  We will check patient's biochemistry profile including, lipid profile, liver function and renal function. Treatment-related adverse events would be assessed by CTCAE v3.0

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No